CLINICAL TRIAL: NCT01529515
Title: A Randomized, Multicenter, Double-Blind, Relapse Prevention Study of Paliperidone Palmitate 3 Month Formulation for the Treatment of Subjects With Schizophrenia
Brief Title: A Study of Paliperidone Palmitate 3 Month Formulation for the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100717; R092670PSY3012 (Other: Janssen Research & Development, LLC); 2011-004676-11 (EudraCT Number); U1111-1135-1969 (Other: Universal Trial Number)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; R092670; Paliperidone Palmitate; Paliperidone palmitate 3 month formulation (PP3M)
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paliperidone palmitate 3-month (PP3M) (Experimental)
  Interventions: Drug: PP3M 175 mg eq.; Drug: PP3M 263 mg eq.; Drug: PP3M 350 mg eq.; Drug: PP3M 525 mg eq.
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (20% Intralipid emulsion)

INTERVENTIONS:
Drug: PP3M 175 mg eq. — Type= exact number, unit= mg eq., number= 175, form= injection, route= intramuscular use. One injection every three months up to the patient has a relapse event or meet discontinuation criteria.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP3M 263 mg eq. — Type= exact number, unit= mg eq., number= 263, form= injection, route= intramuscular use. One injection every three months up to the patient has a relapse event or meet discontinuation criteria.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP3M 350 mg eq. — Type= exact number, unit= mg eq., number= 350, form= injection, route= intramuscular use. One injection every three months up to the patient has a relapse event or meet discontinuation criteria.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: PP3M 525 mg eq. — Type= exact number, unit= mg eq., number= 525, form= injection, route= intramuscular use. One injection every three months up to the patient has a relapse event or meet discontinuation criteria.
  Arms: Paliperidone palmitate 3-month (PP3M)
Drug: Placebo (20% Intralipid emulsion) — Form= injection, route= intramuscular use. One injection every three months up to the patient has a relapse event or meet discontinuation criteria.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of paliperidone palmitate 3 month formulation (PP3M) compared with placebo in delay of the time to first occurrence of relapse of the symptoms of schizophrenia.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double blind (neither physician nor patient knows the treatment that the patient receives), parallel group (each group of patients will be treated at the same time), placebo-controlled (an inactive substance is compared with a drug to test whether the drug has a real effect in a clinical trial) multicenter study. The study consists of 4 phases: a Screening Phase (up to 3 weeks); a 17-week flexible dose open-label Transition Phase (open-label phase means that all people know the identity of the intervention); a 12-week fixed dose open-label Maintenance Phase; and a randomized, double-blind, fixed dose, placebo-controlled relapse prevention phase (referred to as the Double-blind Phase). Patients who meet specific stabilization criteria will enter the Double-blind Phase at Week 29. Patients will be randomly assigned, in a 1:1 ratio, to receive either a fixed dose of PP3M or placebo. The Double-blind Phase will be of variable duration; patients will remain in the study until they experience a relapse event or meet discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia for more than 1 year
* A total score in the Positive and Negative Syndrome Scale (PANSS) < 120
* Signed informed consent
* Women must not be pregnant, breastfeeding, and if capable of pregnancy must practice an effective method of birth control
* Men must agree to use a double-barrier method of birth control
* Be medically stable on the basis of clinical laboratory tests, physical examination, medical history, vital signs, and electrocardiogram (ECG) Exclusion Criteria:
* A diagnosis other than schizophrenia, e.g., dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, primary substance-induced psychotic disorder, dementia-related psychosis
* Relevant history or current presence of any significant or unstable medical condition(s) determined to be clinically significant by the Investigator (ie, obesity, diabetes, heart disease etc)
* A diagnosis of substance dependence within 6 months before screening
* History of neuroleptic malignant syndrome (NMS) or tardive dyskinesia
* Clozapine use in the last 2 months when used for treatment-resistant or treatment-refractory illness
* Clinically significant findings in biochemistry, hematology, ECG or urinalysis results
* Any other disease or condition that, in the opinion of the investigator, would make participation not in the best interest of the patient or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (15):
  - Little Rock, Arkansas
  - San Fran Cisco, California
  - Washington D.C., District of Columbia
  - Lauderhill, Florida
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Topeka, Kansas
  - Baltimore, Maryland
  - Flowood, Mississippi
  - Marlton, New Jersey
  - Cedarhurst, New York
  - Oklahoma City, Oklahoma
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Medellín
  - Pereira
- Malaysia (3):
  - Johor Bahru
  - Kuala Lumpur
  - Tanjong Rambutan
- Mexico (5):
  - Guadajalara
  - Mexico City
  - Monterrey
  - San Luis Potosí City
  - Zapopan
- Romania (5):
  - Arad
  - Craiova
  - Iași
  - Sibiu
  - Tg Mures
- South Korea (4):
  - Deajun
  - Gyeongsangnam-Do
  - Incheon
  - Seongnam
- Turkey (Türkiye) (2):
  - Diyarbakır
  - Sakarya
- Ukraine (15):
  - Donetsk
  - Evpatoriya
  - Hlevakha
  - Ivano-Frankivsk
  - Kerch
  - Kharkiv
  - Kherson
  - Kiev
  - Lviv
  - Odesa
  - Poltava
  - Smila
  - Ternopil
  - Uzhhorod
  - Vinnitsa

REFERENCES:
- [Derived] Mathews M, Gopal S, Singh A, Nuamah I, Pungor K, Tan W, Soares B, Kim E, Savitz AJ. Comparison of Relapse Prevention with 3 Different Paliperidone Formulations in Patients with Schizophrenia Continuing versus Discontinuing Active Antipsychotic Treatment: A Post-Hoc Analysis of 3 Similarly Designed Randomized Studies. Neuropsychiatr Dis Treat. 2020 Jun 19;16:1533-1542. doi: 10.2147/NDT.S221242. eCollection 2020. PMID 32606705
- [Derived] Savitz AJ, Xu H, Gopal S, Nuamah I, Mathews M, Soares B. Efficacy and safety of paliperidone palmitate 3-month formulation in Latin American patients with schizophrenia: A subgroup analysis of data from two large phase 3 randomized, double-blind studies. Braz J Psychiatry. 2019 Nov-Dec;41(6):499-510. doi: 10.1590/1516-4446-2018-0153. PMID 30994855
- [Derived] Weiden PJ, Kim E, Bermak J, Turkoz I, Gopal S, Berwaerts J. Does Half-Life Matter After Antipsychotic Discontinuation? A Relapse Comparison in Schizophrenia With 3 Different Formulations of Paliperidone. J Clin Psychiatry. 2017 Jul;78(7):e813-e820. doi: 10.4088/JCP.16m11308. PMID 28640988
- [Derived] Magnusson MO, Samtani MN, Plan EL, Jonsson EN, Rossenu S, Vermeulen A, Russu A. Population Pharmacokinetics of a Novel Once-Every 3 Months Intramuscular Formulation of Paliperidone Palmitate in Patients with Schizophrenia. Clin Pharmacokinet. 2017 Apr;56(4):421-433. doi: 10.1007/s40262-016-0459-3. PMID 27743205
- [Derived] Gopal S, Vermeulen A, Nandy P, Ravenstijn P, Nuamah I, Buron Vidal JA, Berwaerts J, Savitz A, Hough D, Samtani MN. Practical guidance for dosing and switching from paliperidone palmitate 1 monthly to 3 monthly formulation in schizophrenia. Curr Med Res Opin. 2015 Nov;31(11):2043-54. doi: 10.1185/03007995.2015.1085849. Epub 2015 Oct 2. PMID 26306819
- [Derived] Berwaerts J, Liu Y, Gopal S, Nuamah I, Xu H, Savitz A, Coppola D, Schotte A, Remmerie B, Maruta N, Hough DW. Efficacy and Safety of the 3-Month Formulation of Paliperidone Palmitate vs Placebo for Relapse Prevention of Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Aug;72(8):830-9. doi: 10.1001/jamapsychiatry.2015.0241. PMID 25820612

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 509 participants were enrolled in to the study and 506 participants were entered the Open-label Transition and received at least one dose of study drug (PP1M). 2 participants were enrolled but not received study drug and 1 participant was screen failure.
Groups:
- Open-Label Transition Phase: Paliperidone Palmitate 1-Month: Paliperidone palmitate intramuscular (IM) injection was administered at a dose of 150 milligram equivalents (mg eq) on Day 1, 100 mg eq on Day 8, flexible dose (50, 75, 100, or 150 mg eq) on Day 36 and 64, and on Day 92 same dose as on Day 64.
- Open-Label Maintenance Phase: Paliperidone Palmitate 3-Month: Paliperidone palmitate intramuscular (IM) injection was administered at a dose of 3.5-fold multiple of the PP1M dose received on Day 92 during the Transition Phase.
- Double-Blind Phase: Placebo: Matching placebo [20 percent (%) Intralipid solution] was administered intramuscular (IM) injection every 12 weeks up to participants had a relapse event or met discontinuation criteria.
- Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M): Paliperidone palmitate was administered at a dose of 175, 263, 350, or 525 milligram equivalents (mg eq) intramuscular (IM) injection every 12 weeks up to participants had a relapse event or met discontinuation criteria. Participants received the same dose of study agent that was administered on Day 120 of the Maintenance Phase.
Period: TRANSITION PHASE
Arm/Group | Open-Label Transition Phase: Paliperidone Palmitate 1-Month | Open-Label Maintenance Phase: Paliperidone Palmitate 3-Month | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Started | 506 | 0 | 0 | 0
Completed | 379 | 0 | 0 | 0
Not Completed | 127 | 0 | 0 | 0
Not completed — Adverse Event | 16 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 19 | 0 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 51 | 0 | 0 | 0
Not completed — Failed Maintenance Phase Criteria | 8 | 0 | 0 | 0
Not completed — Other | 9 | 0 | 0 | 0
Period: MAINTENANCE PHASE
Arm/Group | Open-Label Transition Phase: Paliperidone Palmitate 1-Month | Open-Label Maintenance Phase: Paliperidone Palmitate 3-Month | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Started | 0 | 379 | 0 | 0
Completed | 0 | 305 | 0 | 0
Not Completed | 0 | 74 | 0 | 0
Not completed — Adverse Event | 0 | 10 | 0 | 0
Not completed — Lack of Efficacy | 0 | 9 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 0 | 0
Not completed — Protocol Violation | 0 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 15 | 0 | 0
Not completed — Failed Randomization Criteria | 0 | 13 | 0 | 0
Not completed — Other | 0 | 10 | 0 | 0
Period: DOUBLE BLIND PHASE
Arm/Group | Open-Label Transition Phase: Paliperidone Palmitate 1-Month | Open-Label Maintenance Phase: Paliperidone Palmitate 3-Month | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Started | 0 | 0 | 145 | 160
Completed | 0 | 0 | 122 | 148
Not Completed | 0 | 0 | 23 | 12
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 10 | 7
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M) | Total
Number analyzed (Participants) | 145 | 160 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.16) | 37.1 (10.87) | 37.8 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 42 | 77
  Male | 110 | 118 | 228
Region of Enrollment [Number; unit: participants]
  Colombia | 12 | 13 | 25
  Malaysia | 11 | 12 | 23
  Mexico | 10 | 8 | 18
  Romania | 14 | 13 | 27
  South Korea | 4 | 2 | 6
  Turkey | 5 | 6 | 11
  Ukraine | 63 | 74 | 137
  United States | 26 | 32 | 58

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse During the Double-Blind Phase
Description: Time to relapse defined as the time between participant randomization into the double blind Phase and the first documentation of a relapse event. Median time to relapse was estimated by the Kaplan-Meier method.
Time Frame: Approximately Week 60
Population: The intent-to-treat (ITT) double blind (DB) population included all participants who were randomly assigned to treatment during the Double-blind Phase and received at least one dose of Double-blind study agent.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Number analyzed (Participants) | 145 | 160
Days | 395.0 [274.0 to NA] — The NA in the context of the upper limit of a 95% Confidence Interval means "infinity". | NA [NA to NA] — Median time to relapse could not be estimated due to insufficient number of relapses observed in this treatment group.

2. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) (Total Score) From Baseline to Endpoint in the Double-Blind Phase
Description: The PANSS provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items). Each item is rated 1 (absent) to 7 (extreme). The total score ranging from 30 to 210. Higher scores indicate more severe neuropsychiatric symptoms of schizophrenia.
Time Frame: Baseline (Day 1 prior to randomization) and Endpoint (Approximately Week 60)
Population: Intent-to-treat (ITT) double blind (DB) population included all participants who were randomly assigned to treatment during DB Phase and received at least 1 dose of DB study agent. Missing data was imputed using LOCF method. Here "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Number analyzed (Participants) | 142 | 159
Units on a Scale
  Baseline | 54.3 (9.20) | 54.8 (9.96)
  Change at Endpoint (Approximately Week 60) | 6.7 (14.40) | -0.5 (8.36)

3. Secondary Outcome: Change in Clinical Global Impression Severity (CGI-S) Scale From Baseline to Endpoint in the Double-Blind Phase
Description: The CGI-S rating scale is used to rate the severity of a participant's overall clinical condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe).
Time Frame: Baseline (Day 1 prior to randomization) and Endpoint (Approximately Week 60)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Number analyzed (Participants) | 142 | 159
Units on a Scale
  Baseline | 2.8 (0.65) | 2.7 (0.68)
  Change at Endpoint (Approximately Week 60) | 0.4 (0.87) | 0.1 (0.60)

4. Secondary Outcome: Change in Personal and Social Performance (PSP) Scale From Baseline to Endpoint in the Double-Blind Phase
Description: The PSP scale measures personal and social functioning in the domains of: a) Socially useful activities, b) Personal and social relationships, c) Self-care, and d) Disturbing and aggressive behavior. The results of the assessment were converted to a numerical score which ranges from 1 to 100. A score lying between 71 and 100 indicates a mild degree of dysfunction; scores between 31 and 70 indicate varying degrees of difficulty, and a participant with a score of <=30 had functioning so poor that he or she required intensive supervision.
Time Frame: Baseline (Day 1 prior to randomization) and Endpoint (Approximately Week 60)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Number analyzed (Participants) | 142 | 157
Units on a Scale
  Baseline | 68.5 (8.93) | 68.9 (9.34)
  Change at Endpoint (Approximately Week 60) | -4.2 (9.70) | -0.5 (6.63)

ADVERSE EVENTS:
Time Frame: Up to Week 92
Groups:
- Open-Label Phase: PP1M + PP3M: PP1M= Paliperidone Palmitate 1 Month and PP3M= Paliperidone Palmitate 3 Month. Open-Label Transition Phase: Paliperidone palmitate intramuscular (IM) injection was administered at a dose of 150 milligram equivalents (mg eq) on Day 1, 100 mg eq on Day 8, flexible dose (50, 75, 100, or 150 mg eq) on Day 36 and 64, and on Day 92 same dose as on Day 64. Open-Label Maintenance Phase: Paliperidone palmitate intramuscular (IM) injection was administered at a dose of 3.5-fold multiple of the PP1M dose received on Day 92 during the Transition Phase.
Arm/Group | Open-Label Phase: PP1M + PP3M | Double-Blind Phase: Placebo | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M)
Serious Adverse Events (participants affected / at risk) | 33/506 | 15/145 | 4/160
Other Adverse Events (participants affected / at risk) | 317/506 | 77/145 | 98/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Phase: PP1M + PP3M (N=506) | Double-Blind Phase: Placebo (N=145) | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M) (N=160)
Gastritis Erosive (Gastrointestinal disorders) | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 1 | 0 | 0
Transaminases Increased (Investigations) | 0 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Hallucination, Auditory (Psychiatric disorders) | 2 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 9 | 0 | 0
Schizophrenia (Psychiatric disorders) | 12 | 11 | 1
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 | 0 | 1
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 2
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Phase: PP1M + PP3M (N=506) | Double-Blind Phase: Placebo (N=145) | Double-Blind Phase: Paliperidone Palmitate 3-Month (PP3M) (N=160)
Injection Site Pain (General disorders) | 44 | 0 | 2
Nasopharyngitis (Infections and infestations) | 14 | 2 | 9
Weight Decreased (Investigations) | 8 | 11 | 2
Weight Increased (Investigations) | 51 | 5 | 14
Headache (Nervous system disorders) | 33 | 6 | 14
Anxiety (Psychiatric disorders) | 43 | 15 | 13
Insomnia (Psychiatric disorders) | 50 | 17 | 11
Schizophrenia (Psychiatric disorders) | 4 | 8 | 1
Nausea (Gastrointestinal disorders) | 11 | 0 | 2
Fatigue (General disorders) | 13 | 0 | 2
Injection Site Swelling (General disorders) | 11 | 0 | 1
Irritability (General disorders) | 6 | 3 | 1
Influenza (Infections and infestations) | 5 | 3 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 3 | 6
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 5
Blood Glucose Increased (Investigations) | 0 | 3 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Akathisia (Nervous system disorders) | 17 | 1 | 7
Somnolence (Nervous system disorders) | 15 | 0 | 1
Tremor (Nervous system disorders) | 12 | 0 | 2
Agitation (Psychiatric disorders) | 8 | 3 | 2
Suicidal Ideation (Psychiatric disorders) | 13 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. if requested in writing, such publication will be withheld for up to an additional 60 days.